CLINICAL TRIAL: NCT04307810
Title: Parental Expectation for Their Child Behavior in a Group of Children With Primary Dentition During Their First Dental Examination
Brief Title: Parent Predicting of Their Child Behavior During Their First Dental Examination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Alsayed Mohamed Saleh, principal investigator, Cairo University
Other Study IDs: child behavior expectation
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the parental expectation for their child behavior in a group of children with primary dentition during their first dental examination

DETAILED DESCRIPTION:
Assessment of children based on their behavior is one of the most important skills for a pediatric dentist. The major aspect of child management in the dental care is managing dental anxiety and fear as it is considered to be the main barrier for successful completion of dental treatment.

Dental anxiety is a common problem which develops mostly in childhood and adolescence. It can have major implications for the child, dental team, and dental services. Providing treatment for the child with dental anxiety can be time-consuming, costly, and demanding for the clinician.

Previous studies have shown that a majority of children with dental anxiety present behavior management problems (BMP) in dental treatment situations. Evaluating a child's level of anxiety before pediatric treatment is the key, since this anxiety is closely related to their behavior during dental visits. Therefore, predicting the behavior is a basic requirement to reduce child's negative attitude during treatment.

Many behavior rating scales are available to assess and evaluate the behavior of a child on each dental visit. Frankl et al classified child's behavior into four groups according to the child's attitude and cooperation or lack of cooperation during dental treatment. This classification is known as Frankl behavior rating scale, which is one of the most reliable tools developed for behavior rating of children in dental sittings.

ELIGIBILITY:
Inclusion Criteria:

1. Child with Primary dentition
2. First dental visit.
3. Parents of children who agree to fill the questionnaire.

Exclusion Criteria:

1. Child with dental emergency
2. Child with psychological problem
3. Child with chronic illness

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — children with primary dentition
Study Population: children with primary dentition
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Parental expectation for their child behavior | 1 year
  Each parent or caregiver will be asked to fill a questionnaire which includes multiple behavior and actions exhibited by the parents and according to their answers will determine the positive behavior of child

SECONDARY OUTCOMES:
Child behavior | 1 year
  The behavior of the child during his first dental visit will be monitored and videotaped then analyzed in relation to the answers and it well be Measured by using frankl scale.:
  1. _ _ Definitely negative. Refusal of treatment, forceful crying, fearfulness, or any other overt evidence of extreme negativism.
  2. _ Negative. Reluctance to accept treatment, uncooperative, some evidence of negative attitude but not pronounced (sullen, withdrawn).
  3. + Positive. Acceptance of treatment; cautious behavior at times; willingness to comply with the dentist, at times with reservation, but patient follows the dentist's directions cooperatively.
  4. ++ Definitely positive. Good rapport with the dentist, interest in the dental procedures, laughter and enjoyment.